CLINICAL TRIAL: NCT05831930
Title: Radiotherapy Combined With Nitozumab and Sinilimab in the Treatment of Locally Advanced Unresectable Platinum Intolerant Head and Neck Squamous Cell Carcinoma： an Open-label Single-arm, Phase II Trial
Brief Title: The Effect of Nitozumab in the Treatment of Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yangkun Luo, Study Director, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCHEC-02-2023-013
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: Nituozumab

INTERVENTIONS:
Drug: Nituozumab — Nituozumab injection 200mg, administered once a week on the first day, with a duration of at least 60 minutes for a total of 7 times

SUMMARY:
For patients with locally advanced head and neck tumors who are over 70 years old, have PS>2, have hearing impairment, renal dysfunction, or have neuropathy greater than grade 1 that is intolerant to cisplatin, radiotherapy alone or combined with EGFR monoclonal antibody radiotherapy should be chosen. The purpose of this study is to demonstrate the superior efficacy of Nitozumab and Sinilimab when added to radiotherapy in the treatment of high-risk participants with resected locally advanced squamous cell carcinoma of the head and neck (LA SCCHN) who are ineligible to receive cisplatin-based chemoradiation concurrently.

ELIGIBILITY:
Inclusion Criteria:

1.18 years old or above; 2.The subject is a newly diagnosed head and neck squamous cell carcinoma patient who has been confirmed by histopathology or cytology to have stage III-IVB head and neck squamous cell carcinoma (including oral cancer, oropharyngeal cancer, laryngeal cancer, and hypopharyngeal cancer); 3.Tumor tissue samples with positive or weakly positive EGFR immunohistochemistry or FISH detection, i.e. EGFR 2+and EGFR 3+; 4.Locally advanced patients who are not suitable for surgery (referring to patients whose physical conditions do not allow, who refuse surgery due to various reasons, or whose tumor load is too large to be removed), as well as patients with recurrence and metastasis; 5.CPS≥1 6.Absolute contraindications for the use of cisplatin: ECOG ≥ 3 points, creatinine clearance rate<50ml/min, previous hearing impairment or tinnitus ≥ grade 2, grade 2 neuropathy, allergies to drugs containing platinum or mannitol, cardiovascular and respiratory complications, pregnancy, lactation, HIV/AIDS: CD4 count<200/ μ l。 Relative contraindications not suitable for the use of cisplatin: ECOG=2, age>70 years old, creatinine clearance rate 50-60ml/min, previous hearing impairment or tinnitus ≥ 1, grade 1 neuropathy, bone marrow, liver and respiratory dysfunction ≥ 2, Child Pugh score=B, cardiovascular diseases, including hypertension, unstable heart disease, diabetes and repeated lung infections, HIV/AIDS: CD4 count<350/ μ l. Weight loss ≥ 20%, while using nephrotoxic drugs.

7.According to the RECIST 1.1 standard, there is at least one measurable and evaluable target lesion; 8.ECOG score 0-1; 9.The expected survival period exceeds 3 months; 10.Female patients of childbearing age must undergo a negative urine pregnancy test before the start of the study.

Exclusion Criteria:

1. Patients without contraindications for platinum use;
2. Previously received treatment with anti PD-1, anti PD-L1, or any other immune checkpoint inhibitor;
3. Previously received targeted therapy such as EGFR monoclonal antibodies or EGFR tyrosine kinase inhibitors;
4. Participated in other interventional clinical trials within 30 days prior to screening;
5. Other malignant tumors have occurred or are currently suffering from within 5 years, except for cured cervical carcinoma in situ, gastrointestinal intramucosal cancer, breast cancer, skin cancer other than melanoma, and superficial bladder tumor;
6. Active autoimmune diseases that may worsen during immunotherapy;
7. A history of immunodeficiency, including HIV testing positive, active viral hepatitis, tuberculosis, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
8. Inoculate with live vaccine within 30 days of administration.
9. Perform major or planned surgery within 90 days prior to the first administration of the investigational drug;
10. Pregnant (confirmed by blood or urine HCG testing) or lactating women, or subjects of childbearing age who are unwilling or unable to take effective contraceptive measures (applicable to both male and female subjects) until at least 6 months after the last trial treatment;
11. Individuals who are allergic to the use of drugs or their components in this protocol;
12. Those who are unwilling to participate in this study or unable to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 2 years
  The rate of patient complete remission

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China